CLINICAL TRIAL: NCT06856226
Title: Natural History Study to Determine Drug Metabolism Phenotype and Appropriate Germline Source DNA in Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplant
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001796; 001796-C
Record Dates: First submitted 2025-03-01; First posted 2025-03-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12-17

CONDITIONS: Leukemia; Lymphoma; Hematologic Malignancy
Keywords: Allogeneic Transplant; Hematopoietic Cell Transplant; Bone Marrow Transplant; peripheral blood transplant; Chimerism
MeSH Terms: conditions — Leukemia; Lymphoma; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Participants undergoing allogeneic HSCT and donors
  Interventions: Other: Arm 1

INTERVENTIONS:
Other: Arm 1 — Short tandem repeat (STR) analysis from genomic DNA extracted from biospecimens.

SUMMARY:
Background:

After an allogeneic hematopoietic stem cell transplant (HSCT), the donor genome is found in the recipient s circulation and tissues.

Post-HSCT recipients may receive a medication in which the dosing needs to be adjusted based on genetic variation.

While genes in donor genome may influence dosing and administration of some agents, the majority of established gene-drug pairs in pharmacogenetics are related to expression of metabolic or transporting enzymes located in recipients tissues, often the liver.

Determining which genetic variants influence drug disposition in HSCT recipients is complicated by chimerism in samples that are routinely collected for determining genotype. However, chimerism in tissues is poorly studied in this patient population.

Objectives:

To determine the most reliable host genomic source for pharmacogenetic testing in participants that have received allogeneic HSCT.

Eligibility:

People ages 18 years and older who are enrolled on a clinical trial at the NIH Clinical Center under which they will donate or receive an allogeneic HSCT.

Design:

DNA is collected prior to HSCT and for two years after HSCT.

Blood will be collected and skin fibroblast cell lines will be established prior to HSCT to serve as a reference genome.

Blood, buccal cells, skin, and hair will be monitored for the development of mixed chimerism via detection of short tandem repeats. Liver biopsies will be collected from participants undergoing hepatic surgery.

Pharmacoscan arrays will be conducted to determine which samples are useful for pharmacogenetic testing in participants who receive allogeneic HSCT.

A probe drug cocktail will be administered pre- and post-HSCT to determine if transplantation alters the metabolic phenotype of liver enzymes.

...

DETAILED DESCRIPTION:
Background:

* After an allogeneic hematopoietic stem cell transplant (HSCT), the donor genome is found in the recipient fs circulation and tissues.
* Post-HSCT recipients may receive a medication in which the dosing needs to be adjusted based on genetic variation.
* While genes in donor genome may influence dosing and administration of some agents, the majority of established gene-drug pairs in pharmacogenetics are related to expression of metabolic or transporting enzymes located in recipients f tissues, often the liver.
* Determining which genetic variants influence drug disposition in HSCT recipients is complicated by chimerism in samples that are routinely collected for determining genotype. However, chimerism in tissues is poorly studied in this patient population.

Primary Objective:

-To determine the most reliable host genomic source for pharmacogenetic testing in participants that have received allogeneic HSCT.

Eligibility:

* Age >=18 years
* Must be enrolled on a clinical trial at the NIH Clinical Center under which they will donate or receive an allogeneic HSCT

Design:

* DNA is collected prior to HSCT and for two years after HSCT.
* Blood will be collected and skin fibroblast cell lines will be established prior to HSCT to serve as a reference genome.
* Blood, buccal cells, skin, and hair will be monitored for the development of mixed chimerism. Liver biopsies will be collected from participants undergoing hepatic surgery.
* Whole genome sequencing with Aldy analysis will be conducted to determine which samples are useful for pharmacogenetic testing in participants who receive allogeneic HSCT.
* A probe drug cocktail will be administered pre- and post-HSCT to determine if transplantation alters the metabolic phenotype of liver enzymes.
* Up to 88 participants will be enrolled.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age >=18 years
* Participants must be enrolled on a clinical trial at the NIH Clinical Center (CC) under which they will donate or receive an allogeneic HSCT. The participant and their donor must enroll together to provide a complete set of samples for analysis.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Donors are not allowed to enroll without a recipient
* Prior allogeneic HSCT
* History of psychiatric disorder which may compromise compliance with protocol requirements.
* Pregnant and lactating individuals

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any gender, any age greater than or equal to 18 years, who will donate or receive an allogeneic HSCT.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
To determine the most reliable host genomic source for pharmacogenetic testing in participants that have received allogeneic hematopoietic stem cell transplant (HSCT) | Pharmacoscan array will be performed within 1 month pre-BM donation in donors and within 1 month pre-HSCT and 12 months post-HSCT in recipients.
  Obtaining genotype for analysis of pharmacogene activity by understanding the degree chimerism in commonly utilized diagnostic samples.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher G Kanakry, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review and/or will involve genomic data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared after completion of the primary endpoint per the data management sharing plan.
Access Criteria: Data may be requested by contacting the Principal Investigator.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001796-C.html